CLINICAL TRIAL: NCT00273104
Title: The Effect of Lifestyle Intervention vs Gastric Bypass on Various Comorbidities
Brief Title: The Effect of Lifestyle Intervention Versus Gastric Bypass on Various Comorbidities in Morbidly Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital of Vestfold (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Jøran Hjelmesæth, Head of Morbid Obesity Centre, The Hospital of Vestfold
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-05175
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Obstructive Sleep Apnea; Diabetes Mellitus; Hypertension
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus; Hypertension | interventions — Bariatric Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bariatric surgery (Active Comparator): Bariatric surgery (gastric bypass) offered to patients after informed consent and shared decision. The surgical procedure was performed at Vestfold Hospital Trust by experienced bariatric surgeons.
  Interventions: Procedure: Bariatric surgery
- Intensive lifestyle intervention (Active Comparator): Intensive lifestyle intervention (1-year endurance) at a rehabilitation centre. The intervention consisted of motivation for behaviour change including calorie restriction and increased physical activity.
  Interventions: Behavioral: Intensive lifestyle intervention

INTERVENTIONS:
Procedure: Bariatric surgery — Bariatric surgery as a part of public health service offered treatment seeking morbidly obese patients.
  Arms: Bariatric surgery
Behavioral: Intensive lifestyle intervention — Intensive lifestyle intervention as a part of public health service offered treatment seeking morbidly obese patients.
  Arms: Intensive lifestyle intervention

SUMMARY:
This follow up study (>1 year) aims to compare the effects of lifestyle intervention and gastric by pass surgery on various comorbidities associated with morbid obesity.

DETAILED DESCRIPTION:
Not addressed

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patients

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2005-12; Primary Completion 2012-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Improvement of co-morbidities | 1-year after treatment start
  1-year comparative nonrandomized controlled trial

SECONDARY OUTCOMES:
Safety issues | 1-year
  Surgical complications and serious adverse events in both groups as published

CONTACTS AND LOCATIONS:
Overall Officials: Jøran Hjelmesæth, MD PhD, Principal Investigator — Hospital of Vestfold
Locations (1):
- Hospital in Vestfold, Tønsberg, Norway

REFERENCES:
- [Derived] Gabrielsen AM, Omland T, Brokner M, Fredheim JM, Jordan J, Lehmann S, Lund MB, Hjelmesaeth J, Hofso D. The effect of surgical and non-surgical weight loss on N-terminal pro-B-type natriuretic peptide and its relation to obstructive sleep apnea and pulmonary function. BMC Res Notes. 2016 Sep 13;9(1):440. doi: 10.1186/s13104-016-2241-x. PMID 27619215
- [Derived] Hofso D, Birkeland KI, Holst JJ, Bollerslev J, Sandbu R, Roislien J, Hjelmesaeth J. Gastric bypass surgery has a weight-loss independent effect on post-challenge serum glucose levels. Diabetol Metab Syndr. 2015 Aug 22;7:69. doi: 10.1186/s13098-015-0066-8. eCollection 2015. PMID 26300987
- [Derived] Gabrielsen AM, Lund MB, Kongerud J, Viken KE, Roislien J, Hjelmesaeth J, Hofso D. Pulmonary function and blood gases after gastric bypass and lifestyle intervention: a comparative study. Clin Obes. 2013 Oct;3(5):117-23. doi: 10.1111/cob.12024. Epub 2013 Jul 8. PMID 25586626
- [Derived] Karlsen TI, Lund RS, Roislien J, Tonstad S, Natvig GK, Sandbu R, Hjelmesaeth J. Health related quality of life after gastric bypass or intensive lifestyle intervention: a controlled clinical study. Health Qual Life Outcomes. 2013 Feb 13;11:17. doi: 10.1186/1477-7525-11-17. PMID 23406190
- [Derived] Nordstrand N, Hertel JK, Hofso D, Sandbu R, Saltvedt E, Roislien J, Os I, Hjelmesaeth J. A controlled clinical trial of the effect of gastric bypass surgery and intensive lifestyle intervention on nocturnal hypertension and the circadian blood pressure rhythm in patients with morbid obesity. Surgery. 2012 May;151(5):674-80. doi: 10.1016/j.surg.2011.12.007. Epub 2012 Jan 18. PMID 22261295
- [Derived] Fredheim JM, Rollheim J, Omland T, Hofso D, Roislien J, Vegsgaard K, Hjelmesaeth J. Type 2 diabetes and pre-diabetes are associated with obstructive sleep apnea in extremely obese subjects: a cross-sectional study. Cardiovasc Diabetol. 2011 Sep 25;10:84. doi: 10.1186/1475-2840-10-84. PMID 21943153
- [Derived] Hofso D, Jenssen T, Bollerslev J, Ueland T, Godang K, Stumvoll M, Sandbu R, Roislien J, Hjelmesaeth J. Beta cell function after weight loss: a clinical trial comparing gastric bypass surgery and intensive lifestyle intervention. Eur J Endocrinol. 2011 Feb;164(2):231-8. doi: 10.1530/EJE-10-0804. Epub 2010 Nov 15. PMID 21078684
- [Derived] Hofso D, Nordstrand N, Johnson LK, Karlsen TI, Hager H, Jenssen T, Bollerslev J, Godang K, Sandbu R, Roislien J, Hjelmesaeth J. Obesity-related cardiovascular risk factors after weight loss: a clinical trial comparing gastric bypass surgery and intensive lifestyle intervention. Eur J Endocrinol. 2010 Nov;163(5):735-45. doi: 10.1530/EJE-10-0514. Epub 2010 Aug 26. PMID 20798226